CLINICAL TRIAL: NCT05692869
Title: A Study to Investigate Continuous Blood Pressure Monitoring Using Traditional Device (ABPM) Versus Novel Devices (Biobeat and Aktiia)
Brief Title: A Study of Continuous Blood Pressure Monitoring in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 18655; H6O-MC-O017 (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-01-12; First posted 2023-01-20 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Healthy
MeSH Terms: interventions — Propranolol; Pseudoephedrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ABPM + Wearable Novel Devices + Propranolol (Experimental): Participants will wear all the devices (ABPM, chest patch device, wrist device and smartwatch device) with propranolol administered orally for 5 days in one of three study periods.
  Interventions: Drug: Propranolol; Device: ABPM and Wearable Novel Devices
- ABPM + Wearable Novel Devices + Pseudoephedrine (Experimental): Participants will wear all the devices (ABPM, chest patch device, wrist device and smartwatch device) with pseudoephedrine administered orally for 5 days in one of three study periods.
  Interventions: Drug: Pseudoephedrine; Device: ABPM and Wearable Novel Devices
- ABPM + Wearable Novel Devices Only (Experimental): Participants will wear all the devices (ABPM, chest patch device, wrist device and smartwatch device) during one of three study periods.
  Interventions: Device: ABPM and Wearable Novel Devices; Other: No Intervention

INTERVENTIONS:
Drug: Propranolol — Administered orally.
  Arms: ABPM + Wearable Novel Devices + Propranolol
Drug: Pseudoephedrine — Administered orally.
  Arms: ABPM + Wearable Novel Devices + Pseudoephedrine
Device: ABPM and Wearable Novel Devices — ABPM and wearable novel devices including chest patch device, wrist device and smartwatch device worn throughout the trial.
Other: No Intervention — No intervention during this period (Control Period)
  Arms: ABPM + Wearable Novel Devices Only

SUMMARY:
The main purpose of this study in healthy participants is to find out whether the traditional ambulatory blood pressure monitor (ABPM) and newer wearable devices (EmbracePlus smartwatch device, Biobeat chest patch device, and Aktiia wrist device) will accurately pick up changes in blood pressure caused by 2 different medications (propranolol and pseudoephedrine). The study will last about 29 days excluding the screening period of 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy males or females
* Have a body mass index (BMI) of 18.0 to 35 kilograms/square meter (kg/m2), inclusive at screening
* Have blood pressure, pulse rate, blood and urine laboratory test results that are acceptable for the study
* Have given written informed consent approved by Lilly and the ethical review board governing the site

Exclusion Criteria:

* Have or used to have health problems that, in the opinion of the doctor, could make it unsafe to participate, or could interfere with understanding the results of the study
* Have history of sensitive skin or chronic skin conditions, like eczema
* Regular use of known drugs of abuse
* Are women who are pregnant or lactating
* Have known allergies to medications used in the study

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2023-04-04 (Actual); Study Completion 2023-04-04 (Actual)

PRIMARY OUTCOMES:
The Mean Change in Systolic Blood Pressure (SBP) Using Chest Patch Device | Baseline through 48 hours
  The Mean Change in SBP Using Chest Patch Device

SECONDARY OUTCOMES:
The Mean Change in SBP Using Wrist Device | Baseline through 48 hours
  The Mean Change in SBP Using Wrist Device
The Mean Change in Diastolic Blood Pressure (DBP) Using Chest Patch Device and Wrist Device | Baseline through 48 hours
  The Mean Change in DBP Using Chest Patch Device and Wrist Device
The Mean Change in SBP Using Chest Patch Device and Wrist Device | Baseline through 120 hours
  The Mean Change in SBP Using Chest Patch Device and Wrist Device
The Mean Change in DBP Using Chest Patch Device and Wrist Device | Baseline through 120 hours
  The Mean Change in DBP Using Chest Patch Device and Wrist Device
The Mean Change in SBP Using Chest Patch Device, Wrist Device and ambulatory blood pressure monitor (ABPM) | Baseline through 48 hours
  The Mean Change in SBP Using Chest Patch Device, Wrist Device and ABPM
The Mean Change in DBP Using Chest Patch Device, Wrist Device and ABPM | Baseline through 48 hours
  The Mean Change in DBP Using Chest Patch Device, Wrist Device and ABPM

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Lilly Centre for Clinical Pharmacology, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No